CLINICAL TRIAL: NCT06791707
Title: Evaluation of Periodontal Health, Salivary Cotinine and S100A8/A9 Levels in Children Exposed to Secondhand Smoking
Brief Title: Evaluation of Periodontal Health, Salivary Cotinine and S100A8/A9 Levels in Children Exposed to Passive Smoking
Status: Active, not recruiting | Type: Observational
Sponsor: Cumhuriyet University (Other)
Collaborators: Sivas Cumhuriyet Universtiy (Unknown)
Responsible Party: Principal Investigator, Arzu Koçkanat, Assistant Professor, Cumhuriyet University
Other Study IDs: CumhuriyetU_ArzuKockanat_002
Record Dates: First submitted 2025-01-20; First posted 2025-01-24 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-01

CONDITIONS: Secondhand Smoke Exposure; Children; Inflamation; Cotinine Levels

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Passive smoking-exposed children: This group consists of children whose family members have smoked at home since the birth of the child.
- Passive smoking-unexposed children: This group consists of children whose family members have not smoked at home since the birth of the child.

SUMMARY:
The periodontal health of children exposed to passive smoking will be evaluated by S100A8 and S100A9 levels.

DETAILED DESCRIPTION:
Periodontal diseases are inflammatory conditions that affect the tissues supporting the teeth and occur through the interaction between dental plaque and the body's defense response. Microbial biofilm interacts with these tissues to trigger an immune response, and this process leads to changes in proteins, immunoglobulins, and inflammatory markers in the body. S100A8 and S100A9 proteins play an important role in the development of inflammation and are usually found in immune cells.

People exposed to passive smoking have a higher risk of developing periodontal disease. This is related to both microbial effects and changes in immune responses.

In this study, salivary levels of S100A8 and S100A9 proteins, which play a role in inflammation, will be evaluated to determine whether passive smoking increases the risk of periodontal disease in children. 146 children who apply to Sivas Cumhuriyet University Faculty of Dentistry for routine treatment will participate in the study. Their parents will be surveyed about demographic information and smoking habits, and children of parents who regularly smoke at home will be considered as passive smokers, while children of non-smoking parents will be considered as controls. Children who meet the inclusion criteria will be asked to spit into sterile polypropylene tubes for 5 minutes. The saliva flow rate (ml/min) will be measured from the obtained saliva samples and the saliva samples will be centrifuged at 6000 rpm for 10 minutes to remove cell debris. The supernatant phase will be transferred to Eppendorf tubes and stored at -80°C until analysis. Salivary cotinine and S100 A8/A9 levels will be measured using ELISA assay kits following the manufacturer's instructions. The periodontal status of the children will be determined by measuring the whole mouth plaque index (PI), gingival index (GI), probing depth (PD), and clinical attachment level (CAL). All measurements will be made with a dental loupe under 3.5 magnification to increase the accuracy of the data. The data obtained will be recorded on periodontal examination forms. All data obtained will be analyzed using SPSS 23.0 software package program (SPSS Inc., Chicago, IL, USA). Shapiro-Wilk test will be used to examine the normality of data distribution, T test and Mann-Whitney U test will be used to determine the differences between the groups in terms of normal and non-normal data, respectively. Correlations will be analyzed using Spearman's correlation analysis and p<0.05 will be considered significant. As a result of the analysis of the data, the effect of passive smoking on periodontal health in children will be evaluated by comparing the periodontal status and salivary S100A8/A9 and cotinine levels in children exposed to passive smoking and those not exposed.

ELIGIBILITY:
Inclusion Criteria:

* Systemically and genetically healthy children

Exclusion Criteria:

* Any medications known to affect defense system and periodontium
* The presence of orthodontic / intraoral appliance

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All children were selected from patients referred to Sivas Cumhuriyet University, Faculty of Dentistry, and Department of Pediatric Dentistry.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-11-19 (Estimated)

PRIMARY OUTCOMES:
Protein marker | Within 1 year
  S100A8/A9 (pg/mL)

SECONDARY OUTCOMES:
Passive smoking measurement | Within 1 year
  Cotinine (ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Koçkanat, Asst.Prof., Study Chair — Cumhuriyet University
Locations (1):
- Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No